CLINICAL TRIAL: NCT06972797
Title: Accuracy of the DentalSegmentator Tool in 3D Slicer Software Compared to Manual Segmentation in Romixes Software in the Evaluation of Unerupted and Impacted Maxillary Canine: An Observational Study
Brief Title: Accuracy of 3D Slicer Software for Automatic Segmentation Versus Manual Segmentation Using Commercial Software to Evaluate Impacted and Unerupted Maxillary Canine: An Observational Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rabab Amin, Assisstant lecturer, Cairo University
Other Study IDs: CairoU_REC IM031839
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Impacted Canines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our research question will be, can automatic segmentation of maxillary impacted and unerupted canine using DentalSegmentator tool in 3D silcer software be as accurate as manual segmentation?

ELIGIBILITY:
Inclusion Criteria:

Age ranges from 8-70y (from 8 to less than15y for unerupted group - from 15 to 70y for impacted group). b. Scans clearly showing unerupted and impacted maxillary canines.

Exclusion Criteria:

1. Scans with artifacts obscuring the area of interest.
2. Scans with fractures or pathological lesions obscuring the area of interest.
3. Image blurring due to patient movement during acquisition which could interfere with image interpretation.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DICOM data will be collected from the data base anonymously
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
3D volume analysis | one year
  Automatic segmentation of impacted canine and volumetric measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university- faculty of dentistry, Cairo, Cairo Governorate, Egypt